General Template

Version Date: October 2014

Subject Identification

Protocol Title: Omega-3 Fatty Acids for MDD with High Inflammation: A

Personalized Approach

Principal Investigator: David Mischoulon, MD, PhD.

Site Principal Investigator:

Description of Subject Population:Overweight adults with major depressive disorder and elevated inflammatory status

#### About this consent form

Please read this form carefully. It tells you important information about a research study. A member of our research team will also talk to you about taking part in this research study. People who agree to take part in research studies are called "subjects." This term will be used throughout this consent form.

Partners HealthCare System is made up of Partners hospitals, health care providers, and researchers. In the rest of this consent form, we refer to the Partners system simply as "Partners."

If you have any questions about the research or about this form, please ask us. Taking part in this research study is up to you. If you decide to take part in this research study, you must sign this form to show that you want to take part. We will give you a signed copy of this form to keep.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### Why is this research study being done?

We are asking you to take part in a research study. Major depression is a common mental disorder that can have a negative impact on people's lives. Despite the availability of numerous therapies, the current treatment of depression for some people is not ideal. Recently, some research has shown that increasing a diet of polyunsaturated fatty acids (PUFAs), such as omega-3 fatty acids, might help treat depression, especially in depressed people who have highly active immune cells.

We are asking you to take part in this study because you suffer from major depression, are overweight, and may have high levels of immune system markers of inflammation in your


Consent Form Title: Consent form v7

IRB Protocol No: 2015P000944

Consent Form Valid Date: 9/27/2017

IRB Expiration Date: 9/28/2018

Sponsor Protocol No: 3.4

Sponsor AME No: N/A

General Template

Version Date: October 2014



blood. If you are currently on medications for your condition, you are either not doing well on your medications or are experiencing intolerable side effects from your medications. For this study, we will ask you to stop taking any current medications prescribed to you by your doctor.

The purpose of this research study is to compare the effects of three different doses of an omega-3 fatty acid dietary supplement, eicosapentaenoic acid (EPA), versus placebo on immune system markers in the blood and on treating the symptoms of major depression. Eicosapentaenoic acid (EPA) is a common omega-3 fatty acid. EPA is available in low dosages in some types of dietary supplements found in health food stores.

This research study will compare EPA to placebo. The placebo looks exactly like EPA but contains no EPA. During this study, you may get a placebo instead of EPA. Placebos are used in research studies to see if the results are due to the study drug or due to other reasons.

Nordic Naturals ProEPA Xtra Omega-3 food supplement (EPA) is not approved by the U.S. Food and Drug Administration (FDA) to treat Major Depressive Disorder (MDD) with inflammation. That means we are using the supplement for research use only.

This is a pilot study. Pilot studies are done on a small group of subjects to learn if a larger study would be useful. About 250 subjects will take part in this study at MGH, and about 400 subjects in total will take part in this study.

The National Institutes of Health (NIH) National Center for Complementary and Integrative Health (NCCIH) is paying for this study to be done.

#### How long will I take part in this research study?

It will take you about 12 weeks to complete the study. During this time you will be asked to make approximately 9 study visits to MGH. We will also call you 9 times during the study. At the conclusion of the study, you will be offered 3 months of free follow up care with one of the study physicians.

#### What will happen in this research study?

If you decide to take part in this study, you will be asked to stop taking any current medications. After a two to five-week period of not taking your usual medications, you will receive study medication for 12 weeks. You will also undergo standard psychological assessments to monitor your progress. Blood samples will also be collected six times during this study, twice to determine your eligibility to take part in the study, and 4 times to measure changes in immune markers


General Template Version Date: October 2014

| Subject Identification |
|------------------------|

The procedures in this research study are research-related only. Research-related procedures would not be performed if you did not take part in this study.

We will assign you by chance (like a coin toss) to the EPA enriched omega-3-fatty acid preparation group or the placebo group. You and the study doctor cannot choose your study group.

You will have a 25% (1 in 4) chance of being assigned to one of the following groups:

- ☐ Group 1 will receive capsules containing an EPA enriched omega-3 fatty acid preparation for a total dose of 1 g/day.
- Group 2 will receive capsules containing an EPA enriched omega-3 fatty acid preparation for a total dose of 2 g/day.
- ☐ Group 3 will receive capsules containing an EPA enriched omega-3 fatty acid preparation for a total dose of 4 g/day.
- ☐ Group 4 will receive capsules containing placebo (an inactive substance).

You and the study doctor won't know which study group you are in, but the study doctor can find out if necessary.

Both EPA enriched omega-3 fatty acid preparation and placebo will be referred to as 'study drug' from here on in the consent form.

#### Initial Visit-Screening Visit 1 (length of visit about 90 minutes)

Once you agree to participate in this study and sign this consent form, you will be screened by the research staff to determine if you are eligible for the study.

The screening visit will take about 90 minutes and will include the following procedures:

- ☐ A brief physical exam, including a neurologic exam, blood pressure, pulse, height, weight, and a review of your medical history;
- ☐ A psychiatric evaluation
- ☐ A urine drug screen
- ☐ A review of medications you are currently taking
- ☐ An assessment of the amount of omega-3 fatty acids you consume in your diet or in supplements
- ☐ About 2 teaspoons of blood will be drawn from a vein in your arm. Your blood will be tested for an immune marker to determine if you have high immune activation and are eligible for the study.
- ☐ You will be given a food diary and asked to complete the diary on at home for the 3 days before the next screening visit. This diary will monitor your daily dietary intake of foods rich in omega-3 fatty acids.


Consent Form Title: Consent form v7

IRB Protocol No: 2015P000944 Consent Form Valid Date: 9/27/2017

IRB Expiration Date: 9/28/2018

Sponsor Protocol No: 3.4 Sponsor AME No: N/A


| Subject Identification |
|------------------------|

The study team will review the screening data and decide if you are eligible for the study. If you meet entry criteria assessed at screening visit 1, you will come in for screening visit 2.

Elements of the screening visits (V1 and V2) may be combined if you prefer due to time or transportation concerns. If you choose to combine V1 and V2, we will decide if you are eligible for the study after you complete all study procedures for both visits.

#### Second Visit-Screening Visit 2 (length of visit about 90 minutes)

After your blood has been tested and we have determined that you have high immune activation, in order to further determine whether you are eligible to continue to participate in this study, the following tests and procedures will be performed:

| | The food diary will be collected and reviewed |
|--------|-----------------------------------------------|
| $\Box$ | Review of your medical and psychiatric histor |

- ☐ Physical examination, including review of prior and current medications
- About 9 teaspoons of blood will be drawn from a vein in your arm for routine laboratory tests. These tests will screen for medical conditions that may cause depressive symptoms and also screen for pregnancy. A urine sample will be collected to test for the presence of illegal drugs.
- ☐ Electrocardiogram (EKG): This test records the electrical charges that flow through your heart that stimulate it to beat. You will be asked to lie still and relax during the test. A number of wires will be attached with sticky paper to your legs, arms and chest. These wires will be connected to the EKG machine. The machine will record the activity of your heart while you lie still for about 1 minute.

You will be asked to participate in psychological assessments at every visit. We will ask you questions to evaluate your mental health. On average, we think it should take about 30 minutes to complete these assessments. You will be asked to respond to questions about your mental illness, substance abuse, and sexual history. If you feel uncomfortable or embarrassed about answering any question, you may skip it. The questionnaire will be labeled with a unique study number in order to protect your privacy.

If you feel uncomfortable answering any of the questions that we ask you, you are not required to answer them and the researcher will not insist that you respond.

If you are found to be ineligible for this study during either of the screening visits, the research physician will discuss with you alternative therapies and options available to you. Also a list of other research studies available to you will be provided. However, any data collected from you will be kept until the research study is complete. Later in this consent form we will tell you who will be allowed to receive and use any of this information, if you give your permission by signing this consent form.


Consent Form Title: Consent form v7 IRB Protocol No: 2015P000944


| <br>Subject Identification |
|----------------------------|

#### Washout of Psychiatric Medications

If you are currently on a medicine for psychiatric symptoms (except medicines for sleep or anxiety problems) you will need to have stopped them for at least 2 weeks before your Visit 3. Please review the risks of this washout period in the "What are the risks and possible discomforts from being in this research study?" on pages 8 & 9 of this consent form.

If you are already receiving psychotherapy treatment, the study doctor may wish to contact your current mental health counselor/doctor during the washout period to keep him/her informed about changes in your medication. Do you agree to let us contact your current mental health counselor/doctor?

| ☐ YES | □NO | Initials | Date |
|-------|-----|-------------|------|
| | | <del></del> | |

If later you change your mind, please contact the study doctor.

You should not take other medications throughout the study before discussing them with the study physician. You may continue any ongoing psychotherapy treatment you have been receiving for at least 90 days before taking part in this study. However, you cannot begin a new psychotherapy treatment plan while you are taking part in this study.

#### Visit 3 - Baseline visit (length of visit about 120 minutes)

If you continue to qualify for this study, you will be randomized into one of the four study groups. All groups will be instructed to take four capsules of the study medication (or placebo) every morning and another four capsules every afternoon or evening for a total of 8 capsules per day. You will be asked not to change your routine diet during the treatment period and to advise the researcher if you do.

At this visit the following tests and procedures will be performed:

| 11112 | visit the following tests and procedures will be performed: |
|---|---|
| | Vital signs and weight |
| | Questions to allow the researcher to complete standard psychiatric assessments |
| | Review of any medications you are currently taking and your history of tobacco use |
| | Questionnaires that you will be asked to complete |
| | Urine pregnancy test for women able to become pregnant |
| | About 8 teaspoons of blood will be drawn from a vein in your arm. Your blood will be |
| | tested for PUFA profiles, and immunological testing. |
| | Review of possible side effects of study treatment and medication dosing. |

The baseline IDS-C30 at visit 3 may be administered either by telephone 48 hours prior to the visit or in person during the office visit. You will return to see the researcher every 2 weeks at the end of weeks 2, 4, 6, 8, 10 and 12.

You should not become pregnant during this study because the study drug may be harmful to an embryo or fetus. You will provide a urine sample for pregnancy test at this visit.


Consent Form Title: Consent form v7 IRB Protocol No: 2015P000944


Consent Form Valid Date: 9/27/2017

IRB Expiration Date: 9/28/2018


| <br>Subject Identification |
|----------------------------|

| Treatment Visits - Visits 4. 6. and 8 (length of each visit about 60 minutes) |
|---|
| At these visits the following tests and procedures will be performed: Review of possible side effects of study treatment and medication dosing Review of current medications you are taking Questions to allow the researcher to complete standard psychiatric assessment tests. Questionnaires you will be asked to complete |
| If you are unable to attend your scheduled V4, V6, or V8 appointments, all assessments can be completed over the phone and the study will continue as usual. You will be directed to take pills from your extra blister pack until new study medication can be mailed overnight to you. You will have the opportunity to complete your self-report forms online, or have your self-report forms mailed overnight, along with a return envelope so that you can either mail back or scan in your completed self-report forms. Assessments over the phone may not occur more than two times throughout the study. |
| Treatment Visits - Visits 5 and 7 (length of each visit about 90 minutes) At these visits the following tests and procedures will be performed: □ Vital signs and weight □ Review of possible side effects of study treatment and medication dosing □ Review of current medications you are taking □ Questions to allow the researcher to complete standard psychiatric assessment tests □ Questionnaires you will be asked to complete □ About 8 teaspoons of blood will be drawn from a vein in your arm. Your blood will be tested for PUFA profiles, and immunological testing. |
| Final Visit - Visit 9 (length of visit about 90 minutes) □ Vital signs and weight □ Review of possible side effects of study treatment and medication dosing □ Review of current medications you are taking □ Questions to allow the researcher to complete standard psychiatric assessment tests □ Questionnaires you will be asked to complete □ About 8 teaspoons of blood will be drawn from a vein in your arm. Your blood will be tested for PUFA profiles, and immunological testing. □ A urine pregnancy test will be performed for women able to become pregnant □ Collection of study medication |
| Over the course of the study, we will draw approximately 43 teaspoons of blood. |

At visits 3, 5, 7, and 9, you will need to fast before you get your blood drawn. We will ask you to fast from the midnight prior to your visit until after you get your blood drawn. We will ask you to 

| Consent Form Title: Consent form v7 | | |
|---|---|---|
| IRB Protocol No: 2015P000944 | Consent Form Valid Date: 9/27/2017 | IRB Expiration Date: 9/28/2018 |
| Sponsor Protocol No: 3.4 | Sponsor AME No: N/A | IRB AME No: N/A |

General Template

Version Date: October 2014



not eat any food or drink anything besides coffee, tea, or water until after the blood draw is complete. You can take any normal medications you take every morning as well.

#### Who owns my study information and samples?

If you join this study, you will be donating your samples and study information, and you will not receive any compensation for them. If you withdraw from the study, data and samples that were already collected may still be used for this study.

Your samples, genomic data and health information will be stored and shared with other researchers. The samples and information will be available for any research question, such as research to understand what causes certain diseases (for example heart disease, cancer, or psychiatric disorders), development of new scientific methods, or the study of from where different groups of people may have come. No information that would allow anyone outside our group to identify you personally will be released without your written authorization.

We would like to store some of your sample and health information for future studies related to depression. We will label your samples and health information with a code instead of your name. The key to the code connects your name to your sampled and health information. The study doctor will keep the code in a protected computer.

| j <b>g</b> | | , · |
|------------|-----|-----------------------------------------|
| ☐ YES | □NO | Initials |

Do you agree to let us store your sampled for future research related to depression?

If later you change your mind and want your samples destroyed, please contact the study doctor.

If you decide to stop taking part in the study, we will ask you to make a final study visit. The final study will take about 90 minutes. During this visit we will collect/perform the following:

- 1. Vital signs and weight
- 2. Assessment of adverse events
- 3. Review of concomitant medications
- 4. The study doctor will ask you questions about your mental health
- 5. End of Treatment urine pregnancy test if you are a woman able to become pregnant
- 6. Physical Exam
- 7. Phlebotomy for biomarker samples (same as Visit 3)
- 8. Collection of unused study medication

The study doctor may have to take you out of the study. This may happen because:

- 1. You have a serious negative reaction to the study drug
- 2. The study doctor is concerned about your safety
- 3. Your mental health worsens


Consent Form Title: Consent form v7

IRB Protocol No: 2015P000944

Consent Form Valid Date: 9/27/2017


Sponsor AME No: N/A

IRB Expiration Date: 9/28/2018

IRB AME No: N/A


| Sut | ject Identi | fication | <br> |
|-----|-------------|----------|------|

- 4. You are unable to take the study drugs as instructed
- 5. You become pregnant

Partners has an electronic system that lets your study doctors know if you are admitted to a Partners hospital, or if you visit a Partners hospital Emergency Department. We want to make sure the study doctors know about any possible problems or side effects you experience while you are taking part in the study.

A notation that you are taking part in this research study may be made in your electronic medical record. Information from the research that relates to your general medical care may be included in the record (for example: list of allergies, results of standard blood tests done at the hospital labs).

Please ask your doctor if you have any questions about what information will be included in your electronic medical record.

#### **Future Studies**

Dr. Mischoulon and his colleagues are also interested in long-term follow-up studies. We request your permission to be contacted regarding future studies. The sole purpose of this initial contact would be to determine if you are interested in participating in these follow-up studies. Your refusal for future contact will not affect your participation in this research or future research or treatment at Partners Healthcare Institutions.

| You _ | do | _do not agree to be contacted up to | 5 years after the date | e below to determine i | 1 |
|---|---|---|---|---|---|
| you w | ould like | to participate in follow-up studies. | • | | |
| Subjec | t | | Date | | |

# What are the risks and possible discomforts from being in this research study?

While on this study, you may be at risk for certain side effects. There may be other side effects that we cannot predict. Many side effects go away shortly after omega-3-fatty acids are stopped. Also, your condition may not improve or may worsen while you are taking part in this research study. If you have any side effects during the study, you are encouraged to tell the research staff right away.

During the washout period, when you stop taking your current psychotropic medications, your


| Consent Form Title: Consent form v7 | |
|-------------------------------------|------------------------------------|
| IRB Protocol No: 2015P000944 | Consent Form Valid Date: 9/27/2017 |
| Spansor Protocol No: 3.4 | Sponsor AMF No: |


Subject Identification

depression might get worse. If this happens, tell the study doctor. Also, if you have any side effects during the study, please tell the research staff right away.

Omega-3-fatty acids have some reported risks which are mild to moderate in severity. It is likely (occurs in 10-25 out of 100 of subjects) that you will experience some mild stomach upset. The more moderate risks of nausea, diarrhea, bloating, unpleasant belching, and thinning of the blood (which could result in longer bleeding times when cuts or other abrasions occur) are less likely to occur (1-9 out of 100 of subjects).

As with any drug, an allergic reaction can occur with EPA. Allergic reaction can be mild or serious, and can even result in death in some cases. Common symptoms of an allergic reaction are rash, itching, skin problems, swelling of the face and throat, or trouble breathing. If you think you are having an allergic reaction, call the study doctor right away. If you are having trouble breathing, call 911 immediately.

Placebo is an inactive substance, and should not cause any side effects, except for occasional minor stomach upset.

Washout Period: If you are currently on a medicine for psychiatric symptoms (except medicines for sleep or anxiety problems) you will need to have stopped them for at least 2 weeks before your Visit 3 (described above). This is to ensure that there is no residue in your system before beginning the study treatment. If you are depressed despite being on medication, it is likely that the medication you are taking is not working. However, your symptoms of major depression may worsen during this washout period, including thoughts about hurting yourself. You may also experience symptoms of withdrawal from antidepressants, which can include nausea, vomiting, anorexia, headache, flu-like symptoms, tremors, insomnia, and tension. If you feel depressed (excessively sad), develop any unusual or disturbing symptoms, have thoughts about hurting yourself or others, or if any of the symptoms become unmanageable, please inform your study doctor immediately by calling 617-724-5198 and page Dr. Mischoulon. After hours and on weekends, call the MGH Page Operator at 617-726-2066 and have Dr. Mischoulon paged.

If the study physician determines the risk of withdrawing from your current medication is not in your best interest, your participation will be stopped, and other alternatives will be discussed.

**Blood Draw Risks:** Blood drawing may cause some pain and carries a small risk of bleeding, bruising, or infection at the puncture site. There is also a small risk of fainting.

**Instruments and Clinical Interviews:** The instruments that you will be asked to complete and the clinical interviews that you will receive during the course of this study may cause you to feel upset, bored, or fatigued. If you feel uncomfortable answering any of the questions that we ask you, you are not required to answer them and the researcher will not insist that you respond.


Consent Form Title: Consent form v7

IRB Protocol No: 2015P000944


Consent Form Valid Date: 9/27/2017

IRB Expiration Date: 9/28/2018

IRB AME No: N/A


| Subject Identification |
|------------------------|

**Reproductive Risks:** The effect of EPA on an embryo or fetus (developing baby still in the womb), or on a breastfeeding infant, is unknown and may be harmful. Because of these unknown risks, women cannot take part in this study if they are:

☐ Pregnant

☐ Trying to become pregnant

☐ Breastfeeding

If you are a menopausal woman and have not had a period for the past 12 months or more, you will not need to have a pregnancy test. Also, if you have had any well-documented method of surgical sterilization, you will not need to have a pregnancy test. Methods of surgical sterilization include having had a hysterectomy (removal of the uterus with or without the ovaries), bilateral oophorectomy (removal of both ovaries), a tubal ligation (having your tubes tied), or transvaginal occlusion (plugging the opening of the tubes with a coil). All other female subjects must have a negative pregnancy test before starting the study drug.

If you are a female who is sexually active and able to become pregnant, you must agree to use one of the birth control methods listed below. You must use birth control for the entire study, which is at least 12 weeks long, and for 1 week after your last dose of the study drug.

Acceptable birth control methods for use in this study are: oral contraceptives, barrier methods (such as a condom, female condom, or diaphragm), Depo-Provera, spermicidal jelly (a jelly containing the chemical nonoxynol-9 which kills sperm), and an intrauterine device (IUD).

Please ask the researcher about counseling if you would like more information about preventing pregnancy. If you think that you have gotten pregnant during the study, you must tell the study doctor immediately. Pregnant women will be removed from the study.

If you are a man: the effect of EPA on sperm is not known. To protect against possible side effects, if you are a man you should not get a sexual partner pregnant while taking EPA. You and the study doctor should agree on a method of birth control to use throughout the study.

Please keep the study medicine out of the reach of children or anyone else who may not be able to read or understand the label. Do not let anyone else take the medicine besides you.

Incidental Findings: By participating in this study, you will be evaluated with an electrocardiogram and blood tests to assess your overall well-being. Because of these tests, it is possible that you and the investigator might be made aware of a disease that would otherwise not have been detected at this time. This may result in additional testing being recommended by the investigator that you would otherwise not have had. You will be advised of these findings and it is encouraged that you speak to your doctor about them.

It is possible that the researchers will learn something new during the study about the risks of 

Consent Form Title: Consent form v7

IRB Protocol No: 2015P000944

Consent Form Valid Date: 9/27/2017


Sponsor AME No: N/A

IRB AME No: N/A

IRB AME No: N/A


Subject Identification

being in it. If this happens, they will tell you about it. Then you can decide if you want to continue to be in this study or not. You may be asked to sign a new consent form that includes the new information if you decide to stay in the study.

There may be other risks of EPA that are not known yet. If we learn information from you during this study that indicates an intent to seriously harm others or yourself, we may be required by law to share that information with third parties, including public safety or law enforcement authorities, and may take other precautions to protect against such harm.

#### What are the possible benefits from being in this research study?

You may not benefit from taking part in this study. If you receive EPA, it is possible that your depression symptoms will improve while you are taking it. However, although EPA is not FDA-approved, you could purchase this drug over the counter. You will receive the benefit of having your symptoms evaluated, a physical examination, laboratory evaluations, general health discussions with the study doctor, and help with referrals for additional treatment if needed.

We hope the information learned from this study will benefit other patients with depressive symptoms in the future.

#### What other treatments or procedures are available for my condition?

Your participation in this study is completely voluntary. You have the option to not participate in this research study. You may also stop participating in this study at any time.

There are other treatments available for your depression. These include antidepressant medications such as fluoxetine (Prozac), and psychotherapies (talk therapies), such as cognitive-behavioral therapy (CBT).

# Can I still get medical care within Partners if I don't take part in this research study, or if I stop taking part?

Yes. Your decision won't change the medical care you get within Partners now or in the future. There will be no penalty, and you won't lose any benefits you receive now or have a right to receive.

Taking part in this research study is up to you. You can decide not to take part. If you decide to take part now, you can change your mind and drop out later. We will tell you if we learn new information that could make you change your mind about taking part in this research study.

### What should I do if I want to stop taking part in the study?


Consent Form Title: Consent form v7 IRB Protocol No: 2015P000944


Consent Form Valid Date: 9/27/2017

IRB Expiration Date: 9/28/2018

Sponsor AME No: N/A IRB AME No: N/A




If you take part in this research study, and want to drop out, you should tell us. We will make sure that you stop the study safely. We will also talk to you about follow-up care, if needed.

Also, it is possible that we will have to ask you to drop out of the study before you finish it. If this happens, we will tell you why. We will also help arrange other care for you, if needed.

#### Will I be paid to take part in this research study?

You will receive \$20 for the first screening visit and \$25 for the second screening visit. If you choose to combine these two visits, you will receive \$45 for your time visits. After randomization, participants will receive \$40 for every visit they attend with a fasting blood draw (visits 3, 5, 7, and 9) and \$25 for the visits without fasting blood draws (visits 4, 6, and 8). If you do not finish the study, we will compensate you for the visits you have completed. If you complete all study visits, we will pay you \$280 total. You may be asked to fill out a tax form, including your Social Security or Taxpayer Identification Number and U.S. address, in order to be reimbursed, depending on the amount and method of payment. Some payment methods involve mail coming to your house, which may be seen by others in your household. If you have to drive to come to MGH, you will also be provided with parking vouchers at all visits for the MGH garages.

#### What will I have to pay for if I take part in this research study?

The study drug and all of the tests and procedures that will be done only for the research will be paid for by study funds. Charges for any ongoing or routine medical care you receive outside this study will be billed to you or your insurance company in the usual way. You will be responsible for any deductibles or co-payments required by your insurer for your routine medical care.

# What happens if I am injured as a result of taking part in this research study?

We will offer you the care needed to treat any injury that directly results from taking part in this research study. We reserve the right to bill your insurance company or other third parties, if appropriate, for the care you get for the injury. We will try to have these costs paid for, but you may be responsible for some of them. For example, if the care is billed to your insurer, you will be responsible for payment of any deductibles and co-payments required by your insurer.

Injuries sometimes happen in research even when no one is at fault. There are no plans to pay you or give you other compensation for an injury, should one occur. However, you are not giving up any of your legal rights by signing this form.

If you think you have been injured or have experienced a medical problem as a result of taking 

Consent Form Title: Consent form v7 IRB Protocol No: 2015P000944

Consent Form Valid Date: 9/27/2017

IRB Expiration Date: 9/28/2018


Sponsor AME No: N/A


| <br>Subject Identi | fication |
|--------------------|----------|

part in this research study, tell the person in charge of this study as soon as possible. The researcher's name and phone number are listed in the next section of this consent form.

# If I have questions or concerns about this research study, whom can I call?

You can call us with your questions or concerns. Our telephone numbers are listed below. Ask questions as often as you want.

David Mischoulon, MD, PhD is the person in charge of this research study. You can call him at 617-724-5198, during the hours of 9:00AM and 5:00PM, Monday through Friday. You can page him at 617-726-2066 24 hours a day, 7 days a week. You can also call Lisa Sangermano at 617-724-3673 during the hours of 9:00AM and 5:00PM, Monday through Friday with questions about this research study.

If you have questions about the scheduling of appointments or study visits, call Lisa Sangermano at 617-724-3673.

If you want to speak with someone **not** directly involved in this research study, please contact the Partners Human Research Committee office. You can call them at 857-282-1900.

You can talk to them about:

| Your rights as a research subject |
|-----------------------------------|
| Your concerns about the research |
| A complaint about the research |

Also, if you feel pressured to take part in this research study, or to continue with it, they want to know and can help.

### If I take part in this research study, how will you protect my privacy?

During this research, identifiable information about your health will be collected. In the rest of this section, we refer to this information simply as "health information." In general, under federal law, health information is private. However, there are exceptions to this rule, and you should know who may be able to see, use, and share your health information for research and why they may need to do so.

#### In this study, we may collect health information about you from:

| Past, present, and future medical records |
|---|
| Research procedures, including research office visits, tests, interviews, and |
| questionnaires |

Who may see, use, and share your identifiable health information and why they may need to do so:


| Consent Form Title: Consent form v7 | | |
|---|---|---|
| IRB Protocol No: 2015P000944 | Consent Form Valid Date: 9/27/2017 | IRB Expiration Date: 9/28/2018 |
| Sponsor Protocol No: 3.4 | Sponsor AME No: N/A | IRB AME No: N/A |


| Subject Identification |
|------------------------|

| Partners research staff involved in this study |
|---|
| The sponsor(s) of this study, and the people or groups it hires to help perform this research |
| Other researchers and medical centers that are part of this study and their ethics boards |
| A group that oversees the data (study information) and safety of this research |
| Non-research staff within Partners who need this information to do their jobs (such as for treatment, payment (billing), or health care operations) |
| The Partners ethics board that oversees the research and the Partners research quality improvement programs. |
| People from organizations that provide independent accreditation and oversight of hospitals and research |
| People or groups that we hire to do work for us, such as data storage companies, insurers, and lawyers |
| Federal and state agencies (such as the Food and Drug Administration, the Department of Health and Human Services, the National Institutes of Health, and other US or foreign government bodies that oversee or review research) |
| Public health and safety authorities (for example, if we learn information that could mean harm to you or others, we may need to report this, as required by law) |
| Other: |

Some people or groups who get your health information might not have to follow the same privacy rules that we follow and might use or share your health information without your permission in ways that are not described in this form. For example, we understand that the sponsor of this study may use your health information to perform additional research on various products or conditions, to obtain regulatory approval of its products, to propose new products, and to oversee and improve its products' performance. We share your health information only when we must, and we ask anyone who receives it from us to take measures to protect your privacy. The sponsor has agreed that it will not contact you without your permission and will not use or share your information for any mailing or marketing list. However, once your information is shared outside Partners, we cannot control all the ways that others use or share it and cannot promise that it will remain private.

Because research is an ongoing process, we cannot give you an exact date when we will either destroy or stop using or sharing your health information.

The results of this research study may be published in a medical book or journal, or used to teach others. However, your name or other identifying information will not be used for these purposes without your specific permission.

#### **Your Privacy Rights**


Consent Form Title: Consent form v7 IRB Protocol No: 2015P000944


Consent Form Valid Date: 9/27/2017

IRB Expiration Date: 9/28/2018

IRB AME No: N/A

General Template
Version Date: October 2014

Subject Identification

You have the right **not** to sign this form that allows us to use and share your health information for research; however, if you don't sign it, you can't take part in this research study.

You have the right to withdraw your permission for us to use or share your health information for this research study. If you want to withdraw your permission, you must notify the person in charge of this research study in writing. Once permission is withdrawn, you cannot continue to take part in the study.

If you withdraw your permission, we will not be able to take back information that has already been used or shared with others.

You have the right to see and get a copy of your health information that is used or shared for treatment or for payment. To ask for this information, please contact the person in charge of this research study. You may only get such information after the research is finished.

#### **Email Encryption Preference**

The Partners standard is to send email securely. This requires you to initially set up and activate an account with a password. You can then use the password to access secure emails sent to you from Partners HealthCare. If you prefer, we can send you "unencrypted" email that is not secure and could result in the unauthorized use or disclosure of your information. If you want to receive communications by unencrypted email despite these risks, Partners HealthCare will not be held responsible. Your preference to receive unencrypted email will apply to emails sent to you from research staff in this study ONLY.

Please select one of the following options:

| I consent to receive unencryp | ted emails (please use your initials to indicate your response): |
|---|---|
| Yes: | No: |

#### **Informed Consent and Authorization**

#### Statement of Person Giving Informed Consent and Authorization

| I have read this consent form. |
|---|
| This research study has been explained to me, including risks and possible benefits (if |
| any), other possible treatments or procedures, and other important things about the study. |
| I have had the opportunity to ask questions. |
| I understand the information given to me. |

Signature of Subject:


Consent Form Title: Consent form v7

IRB Protocol No: 2015P000944

Consent Form Valid Date: 9/27/2017


Sponsor AME No: N/A

IRB Expiration Date: 9/28/2018

| Cubicat Identification |
|------------------------|
| Subject Identification |

| General Template<br>Version Date: October 2014 | | Subject Identification |
|---|---|---|
| I give my consent to take part in this research stube used and shared as described above. | dy and agree to | allow my health information to |
| Subject | Date | Time (optional) |
| Signature of Study Doctor or Person ( | Obtaining Co | nsent: |
| ☐ I have explained the research to the study☐ I have answered all questions about this i | - | the best of my ability. |
| Study Doctor or Person Obtaining Consent | Date | Time |
| Subject's Spoken Language Statement of Hospital Medical Interpreter As someone who understands both English and the subject's language, the researcher's presentation given the opportunity to ask questions. | | |
| Hospital Medical Interpreter | Date | Time (optional) |
| OR Statement of Other Individual (Non-Interpre As someone who understands both English and represent that the English version of the consent the subject's own language, and that the subject questions. | the language spo<br>form was preser | nted orally to the subject in |
| Name | Date | Time (optional) |
| Consent Form Version: September 22, 2017 | | |


Consent Form Title: Consent form v7 IRB Protocol No: 2015P000944

Consent Form Valid Date: 9/27/2017

IRB Expiration Date: 9/28/2018

IRB AME No: N/A
